CLINICAL TRIAL: NCT04706234
Title: Prospective Observational Study for the Systematic Assessment of Laryngopharyngeal Function in Patients With Neurodegenerative Diseases
Brief Title: Systematic Assessment of Laryngopharyngeal Function in Patients With Neurodegenerative Diseases
Acronym: FEEMSA
Status: Recruiting | Type: Observational
Sponsor: Kliniken Beelitz GmbH (Other)
Collaborators: University Hospital Muenster (Other); Medical University of Warsaw (Other); Hannover Medical School (Other); University of Ulm (Other); Medical University Innsbruck (Other); University Hospital Carl Gustav Carus (Other); University of Barcelona (Other); Seoul National University Hospital (Other); Gifu University Graduate School of Medicine (Other); University of Bologna (Other); Tel Aviv University (Other); Asklepios Kliniken Hamburg GmbH (Other); Asklepios Fachklinikum Stadtroda (Other); Klinikum Osnabrück (Unknown)
Responsible Party: Principal Investigator, Florin Gandor, MD, Consultant Neurologist, Kliniken Beelitz GmbH
Other Study IDs: S21(a)/2017
Record Dates: First submitted 2021-01-09; First posted 2021-01-12 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Multiple System Atrophy; Parkinson Disease; Progressive Supranuclear Palsy; Motor Neuron Disease; Neurodegenerative Diseases
Keywords: Multiple System Atrophy; Progressive Supranuclear Palsy; Parkinson's disease; Motor Neuron Disease; Neurodegenerative Diseases; Dysphagia; FEES; Laryngeal EMG; Irregular Arytenoid Cartilages Movements; Clinical Biomarker
MeSH Terms: conditions — Multiple System Atrophy; Parkinson Disease; Supranuclear Palsy, Progressive; Motor Neuron Disease; Neurodegenerative Diseases; Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Multiple System Atrophy: Patients diagnosed will probable or possible MSA according to the 2nd criteria for the diagnosis of MSA (Gilman 2008) that received laryngopharyngeal assessment according to the systematic task protocol during FEES (Warnecke et al. 2019).
- progressive supranuclear palsy: Patients diagnosed will probable or possible Progressive Supranuclear Palsy or (PSP) related 4repeat tauopathies according to the Movement Disorders Society diagnostic criteria (Höglinger 2017) that received laryngopharyngeal assessment according to the systematic task protocol during FEES (Warnecke et al. 2019).
- Parkinson Disease: Patients diagnosed will Parkinson's disease according to the Movement Disorders Society diagnostic criteria (Postuma 2015) that received laryngopharyngeal assessment according to the systematic task protocol during FEES (Warnecke et al. 2019).
- Motor Neuron Disease: Patients diagnosed with Motor Neuron Disease that received laryngopharyngeal assessment according to the systematic task protocol during FEES (Warnecke et al. 2019).
- Neurodegenerative Diseases: Patients diagnosed with a neurodegenerative disease not specified above that received laryngopharyngeal assessment according to the systematic task protocol during FEES (Warnecke et al. 2019).

SUMMARY:
This is a non-interventional observational study designed to systematically record the results of routine laryngeal examinations and specific characteristics of dysphagia in patients with neurodegenerative disorders. The results of a fiberoptic / flexible endoscopic evaluation of swallowing (FEES) while performing a structured task protocol will be recorded. If available, laryngeal electromyography (EMG) results will also be recorded. In addition to the examination results, demographic and disease-specific data are collected, and two questionnaires, the Swallowing Disturbance Questionnaire for Parkinson's Disease (SDQ-PD) and the swallowing specific Quality Of Life Questionnaire (SWALQOL), are administered.

DETAILED DESCRIPTION:
Neurodegenerative disorders are associated with a high prevalence of neurogenic dysphagia. Depending on the underlying disease, the prevalence can affect up to 80% of patients. Dysphagia is associated with dehydration, malnutrition, facilitates aspiration pneumonia and thereby determines the prognosis of neurodegenerative diseases. For most of them, dysphagia-associated complications are the leading cause of death.

Multiple system atrophy (MSA) is a sporadic progressive neurodegenerative disorder caused by oligodendroglial aggregation of α-synuclein affecting predominantly the nigrostriatal, olivo-ponto-cerebellar, and autonomic systems,resulting in a clinical presentation of dysautonomia combined with either predominantly parkinsonian (MSA-P) or cerebellar (MSA-C) symptoms of varying severity.In its early stage, the diagnosis of MSA according to the second consensus criteria can be challenging. Therefore, the Movement Disorders Society MSA study group recently addressed the importance of developing valuable diagnostic tools for securing an early diagnosis in patients with MSA not only to estimate disease prognosis but also to early initiate novel, potentially disease-modifying treatments in clinical trials. Despite laryngopharyngeal dysfunction being associated with decreased life expectancy and quality of life, systematic assessment of these functions in MSA is scarce. Previously, an easy-to-implement MSA-FEES task-protocol was suggested to systematically assess laryngopharyngeal function.

A pilot study on 8 patients with MSA not only showed that the task protocol was feasible and well tolerated, but also that laryngopharyngeal symptoms where highly prevalent despite the lack of clinical presentation (Warnecke et. al 2019). Moreover, irregular arytenoid cartilages movements where present in all MSA-patients when performing this task protocol, suggesting this symptom could serve as a clinical marker to identify MSA-patients. Following this pilot study, an observational two center study assessed 57 MSA patients with this protocol and compared findings to an age-matched cohort of PD-patients (Gandor et al. 2020). While only 43.9% of MSA patients had clinical symptoms of laryngeal dysfunction, 93% showed laryngeal abnormalities during FEES performing the task-protocol. 91.2% of MSA-patients showed irregular arytenoid cartilages movements. In contrast, only one PD patient showed laryngeal abnormalities with vocal fold motion impairment, but not irregular arytenoid cartilages movements. This study suggests that irregular arytenoid cartilages movements allow differentiating MSA from PD with a sensitivity of 0.9 and a specificity of 1.0.

4repeat tauopathies (4RT) are caused by an intraneuronal accumulation of 4repeat tau.

4RT, also known as progressive supranuclear palsy (PSP) with all its clinical subtypes, is a rapidly progressive neurodegenerative disease that leads to increasing impairment of cortical and subcortical function in the affected person due to the accumulation of tau protein in the brain (Höglinger 2017). Due to the clinical variability of the presentation, early diagnostic certainty is desirable. Depending on the affected area in the central nervous system, different clinical phenotypes result. The most commonly described and researched entity is Progressive Supranuclear P, also known as Richardson Syndrome, or PSP-RS. Further clinical presentations include a Parkinsonian variant (PSP-P), corticobasal syndrome (PSP-CBS), pure akinesia with gait freezing (PSP-PAGF), speech/language dominant presentations (PSP-SL), frontotemproal dementia variants (PSP-FTD), and cerebellar presentations (PSP-C) (Höglinger 2017).

4RT is also associated with swallowing and speech problems, and aspiration pneumonia is one of the most common causes of death in this disease entity (Tilley 2016). In addition, dystonic dysinnervation of laryngeal muscles can lead to laryngeal motion abnormalities (Panegyres 2007).

Equally, patients with motor neurone disease (MND) are affected by dysphagia early in the disease. In a FEES study by Steven B. Leder and colleagues (2004), which included 17 ALS patients subjectively complaining of dysphagia, fluid aspiration or an increased risk of fluid aspiration was found in almost 60% of cases, regardless of whether the disease initially mainly affected the bulbar musculature or the limb musculature. As the disease progressed, the depth of penetration of fluids into the hypopharynx prior to triggering the swallowing reflex increased, so these patients were advised to thicken fluids. Initially, residues of solid food consistencies were detected in the valleculae, piriform sinus and/or laryngeal inlet in three patients after swallowing. As a result of progressive paresis of the pharyngeal muscles, the residuals increased in the ALS patients examined during the course of the disease. If this disorder pattern was detected, it was advised to reduce the size of the food bolus and to clear the pharynx by swallowing water or reswallowing several times. In a further small case series (n = 11), the FEES showed that dysphagic ALS patients are particularly at risk of penetration/aspiration when swallowing liquids. Penetration and aspiration occur particularly frequently intradeglutitively (D'Ottaviano et al. 2013). A recent publication reports on FEES examinations in 202 ALS patients (w/m 95/107; bulbar/spinal onset 66/136; mean age 64.68 +/- 11.12 years). A close positive correlation with disease severity (measured using the ALSFRS-R) was found for all FEES parameters (leaking, aspiration, residuals), regardless of the three consistencies tested (liquid, semi-solid, solid) (Fattori et al. 2017).

The aim of this FEEMSA trial is to continue recruitment of patients with neurodegenerative diseases and systematically assess laryngopharyngeal function in large cohorts, to categorise the dysphagia phenotypes and better correlate them with the disease subtypes (MSA Parkinson vs cerebellar; PSP variants, MND variants, etc). If available, laryngeal EMG will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of probable or possible multiple system atrophy according to current consensus criteria (Gilman et al. 2008) or
* diagnosis of probable or possible PSP according to the the Movement Disorders Society (MDS) diagnostic criteria (Höglinger et al. 2017) or
* diagnosis of Parkinson's disease according to the MDS diagnostic criteria (Postuma et al 2015)
* Hoehn and Yahr Stage within the range of I-V or
* diagnosis of motor neurone disease or
* diagnosis of a neurodegenerative disease other than specified above

AND underwent laryngopharyngeal assessment according to the systematic task protocol during FEES (Warnecke et al. 2019).

Exclusion Criteria:

- Patients who do not sign the consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited at the participating sites from outpatient's clinics or admitted patients.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
laryngeal movement disorders | 1 day
  occurrence of vocal fold motion impairment, paradoxical vocal fold motion, vocal fold fixation or involuntary irregular arytenoid cartilages movements when assessed with the task-protocol
dysphagia | 1 day
  occurrence of dysphagic symptoms when assessed with the task-protocol

OTHER OUTCOMES:
laryngeal EMG findings | 1 day
  abnormalities recorded on laryngeal EMG showing denervation, dystonic co-activation or myoclonic discharges

CONTACTS AND LOCATIONS:
Overall Officials: Florin Gandor, MD, Principal Investigator — Movement Disorders Hospital Beelitz-Heilstätten, Germany
Locations (16):
- Department of Neurology and Department of ENT, Medical University Innsbruck, Innsbruck, Tyrol, Austria
- Germany (9):
  - Department of Neurology, Medical University of Ulm, Ulm, Baden-Wurttemberg
  - Movement Disorders Hospital - Kliniken Beelitz, Beelitz-Heilstätten, Brandenburg
  - Department of Neurology, Medical School Hannover, Hanover, Lower Saxony
  - Department of Neurology, University Hospital Münster, Münster, North Rhine-Westphalia
  - Department of Neurology, University Hospital Carl Gustav Carus, Dresden, Saxony
  - Department of Neueology Asklepios Klinik Stadtroda, Stadtroda, Thuringia
  - Asklepios Fachklinikum Stadtroda, Stadtroda, Thuringia
  - Asklepios Klinik Barmbek, Hamburg
  - Department of Neurology Asklepios Klinik Barmbek, Hamburg
- Department of Neurology, Movement Disorders Unit, Medical Center Tel Aviv, Tel Aviv, Israel
- IRCCS Istituto delle Scienze Neurologiche, Azienda USL di Bologna, Bologna, Italy
- Department of Neurology, Gifu University Graduate School of Medicine, Gifu, Japan
- Department of Neurology, Medical University Warsaw, Warsaw, Poland
- Department of Neurology SNUCM, Seoul, South Korea
- Unidad de Parkinson y Trastornos del Movimiento Instituto Clínic de Neurociencias, Hospital Clinic de Barcelona, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Warnecke T, Vogel A, Ahring S, Gruber D, Heinze HJ, Dziewas R, Ebersbach G, Gandor F. The Shaking Palsy of the Larynx-Potential Biomarker for Multiple System Atrophy: A Pilot Study and Literature Review. Front Neurol. 2019 Mar 26;10:241. doi: 10.3389/fneur.2019.00241. eCollection 2019. PMID 30972002
- [Background] Gandor F, Vogel A, Claus I, Ahring S, Gruber D, Heinze HJ, Dziewas R, Ebersbach G, Warnecke T. Laryngeal Movement Disorders in Multiple System Atrophy: A Diagnostic Biomarker? Mov Disord. 2020 Dec;35(12):2174-2183. doi: 10.1002/mds.28220. Epub 2020 Aug 5. PMID 32757231
- [Background] Vogel A, Claus I, Ahring S, Gruber D, Haghikia A, Frank U, Dziewas R, Ebersbach G, Gandor F, Warnecke T. Endoscopic Characteristics of Dysphagia in Multiple System Atrophy Compared to Parkinson's Disease. Mov Disord. 2022 Mar;37(3):535-544. doi: 10.1002/mds.28854. Epub 2021 Nov 13. PMID 34773420